CLINICAL TRIAL: NCT00362258
Title: Irbesartan In Hypertensive Diabetic Patients
Brief Title: I PREVENT - Irbesartan In Hypertensive Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0256
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Irbesartan (Aprovel) — Aprovel (150 & 300mg) & CoAprovel (300/12.5mg hydrochlorothiazide) one tablet/day per os.

SUMMARY:
* To evaluate Blood Pressure (BP) reduction to the targeted values (Systolic BP ≤ 130 mmHg and Diastolic BP ≤ 80 mmHg) in hypertensive type 2 diabetic patients.
* To evaluate the benefit of Irbesartan in the reduction of microalbuminuria from baseline (if any at the inclusion visit) in this population.
* To demonstrate the safety of Irbesartan in this population.

ELIGIBILITY:
Inclusion Criteria:

* Proven Hypertensive Type 2 Diabetic Patients with HbA1c > 6% and ≤ 10% (with or without microalbuminuria).
* Newly diagnosed "naïve" hypertensive patients (no prior treatment for hypertension). OR,
* Patients who were receiving antihypertensive agents (maximum two agents, including one diuretic) with blood pressure targets achieved, yet, in the investigator's opinion, those patients would benefit more from switching to the study medication. These patients will undergo a wash out period for not less than 7 days prior to enrollment.

Exclusion Criteria:

* Severe hypertension (SBP ≥ 180 mm Hg or DBP ≥ 110 mm Hg).
* Patients with secondary hypertension.
* Patients with UAE > 200µg / min.
* Patients with HbA1c < 6% or > 10%.
* Significant chronic renal impairment (Serum creatinine > 2.0 mg/dL).
* Significant liver disease as shown by SGPT/SGOT (ALAT/ASAT) > 2.5 times the upper limit of the normal range.
* Currently pregnant or lactating females.
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Any patient who is in need for a combination antihypertensive therapy from the start (from the medical point of view of his/her physician).
* Known hypersensitivity to irbesartan, other ARBs(Angiotensin Receptor Blockers), hydrochlorothiazide, or other thiazide diuretics.
* Patients with malignancy during the past 5 years, known collagen disease or severe cardiac, cerebrovascular or gastric disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Reach blood pressure target in hypertensive diabetic patients i.e. 130/80 mmHg. | During the study conduct

SECONDARY OUTCOMES:
The restoration of urinary albumin excretion (UAE) rate in patients with normoalbuminuria (UAE rate < 20µg / min) | During the study conduct
First detection of overt nephropathy (UAE rate > 200µg / min), in patients with microalbuminuria or at least 30% higher than at baseline value(on at least two consecutive occasions) | During the study conduct
Occurrence of any side effect leading to treatment discontinuation. | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Mosaad I Morsi, MBBCh, MSc, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Cairo, Egypt